CLINICAL TRIAL: NCT03342716
Title: Resolution of Organ Injury in Acute Pancreatitis - RESORP
Acronym: RESORP
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: v11 23 Sept 2019; MR/P008887/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2017-09-29; First posted 2017-11-17 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-02

CONDITIONS: Pancreatitis, Acute
Keywords: Pancreatitis; Multiple Organ Dysfunction Syndrome
MeSH Terms: conditions — Pancreatitis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both DNA and RNA samples taken at baseline, 3 and 36 month visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main cohort: Patients with a clinical or radiological diagnosis of acute pancreatitis (AP)
- Nested cohort: Subgroup of patients with a clinical or radiological diagnosis of acute pancreatitis (AP) who will undergo additional assessments and scans

SUMMARY:
Acute pancreatitis (AP) is inflammation of the pancreas usually triggered by gallstones or drinking excessive alcohol. 80% of people who have an episode of AP will recover without complications. However, 20% will require treatment in high dependency or intensive care for multiple organ dysfunction (AP-MODS). It is known that this negatively affects recovery and can have a lasting effect on health although it is incompletely understood what causes this.

Aim: To recruit 500 patients with acute pancreatitis. Participants will be assessed at recruitment and and again at 3 and 36 months. Recovery of organ function will be serially measured and the presence of novel factors important in recovery assessed.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a common and devastating disease with an annual incidence of 22-30 per 100,000 in the UK. The incidence is increasing. AP is most commonly triggered by gallstones or alcohol excess and has a range of outcomes, from complete resolution to death, with an overall mortality in Scotland of 5.2%. AP is characterised by acute inflammation of the pancreas, which initiates a cascade of inflammatory events throughout the body that can lead to multiple organ dysfunction syndrome (MODS) in approximately 25% of AP patients. Mortality in AP is greatest in those patients who develop MODS, with death rates reported to be up to 28%.

The development of persistent organ failure characterises severe AP (SAP) as defined in the revised Atlanta classification, and is strongly predictive of a fatal outcome. A significant proportion of research has focussed on reducing mortality and morbidity in the first week. As a consequence, it remains to be seen whether the patterns of early organ dysfunction are reflected in the causes of long-term mortality and morbidity.

Recently published data from a retrospective analysis of patients admitted to the Royal Infirmary of Edinburgh with acute pancreatitis has shown that the early development of MODS is associated with an increased mortality rate up to 10 years after the index presentation. This strongly suggests that MODS in acute pancreatitis (AP-MODS) has a persistent and deleterious impact on patients' physiological status, though the exact nature of this pathology remains to be characterised. Recent data has indicated that the severity of the first attack of AP significantly influences the risk of progression to chronic pancreatitis, and therefore subsequent long-term morbidity.

This observational clinical cohort study aims to characterise the nature and extent of the pathophysiological impact of SAP on organ function over the first 3 years following the index event and the long-term deleterious effect of SAP. This will be achieved by prospectively evaluating the pathophysiological consequences of an episode of AP by measuring organ system function in patients recruited during a hospital admission with AP. We will obtain an in-depth assessment of patients' health at presentation, and at 3 months and 36 months after the first episode of AP using markers of organ function and/or disease in the peripheral blood. In a nested cohort within the main study cohort, we will conduct cardiorespiratory evaluation tests (including exercise testing), specialised blood tests of the immune system, tests for precision medicine, and imaging to assess structure and function of key organ systems.

The results of this study will inform the design of future interventions designed to improve the long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

All patients treated at Royal Infirmary Edinburgh with a clinical or radiological diagnosis of acute pancreatitis will be recruited where possible.

For the potential clinical diagnosis of acute pancreatitis an appropriate clinical history based on compatible clinical features, will be required (i.e. abdominal pain, nausea and/or vomiting), supported by the finding of elevated serum amylase greater than 3x the upper limit of the reference range for the laboratory (currently 300 U/L).

For the radiological diagnosis, if applicable, computerised tomography (CT) and/or ultrasound scan (USS) evidence of acute pancreatitis will be accepted.

Exclusion Criteria:

The following exclusion criteria will be adhered to:

i. Patients under the age of 16 years will be excluded from the present study. ii. Prisoners will be excluded from the present study. iii. Patients lacking the capacity to consent will be excluded but can be included if they regain capacity.

Additional exclusions will apply only to those patients being considered for the nested cohort study:

iv. Patients not able to undergo MRI scanning for technical reasons will be excluded (e.g. those with cochlear implants, implanted pacemaker) v. Patients with a known allergy to salbutamol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated at the Royal Infirmary Edinburgh with a clinical or radiological diagnosis of acute pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Annual incidence of new-onset type 3c diabetes mellitis in patients with AP | 66 months
  Do patients that have had AP develop type 3c diabetes mellitis more frequently?
Nested cohort only - difference in the 3 month to 36 month change in pancreatic fibrosis index between participants with AP with MODS and those with AP without MODS | 66 months
  Assess any damage to pancreas at 3 and 36 months and monitor how this changes throughout the course of the trial comparing participants with AP only and those with AP and MODS

SECONDARY OUTCOMES:
Specific gene and promoter sequence variation between participants with AP and AP-MODS | 66 months
  Define any gene and promoter sequence variation between participants with AP and AP-MODS; machine learning approach
miRNA signatures of disease severity and resolution | 66 months
  Comparing patterns of gene expression in mild/moderate/severe cases of AP; machine learning approach
Metabolomic profiling of AP resolution. | 66 months
  Comparing patterns of metabolite expression in mild/moderate/severe cases of AP; machine learning approach
Incidence of premature cellular senescence as a pathological consequence of AP-MODS. | 66 months
  Investigating pathological consequences of AP-MODS compared to AP without MODS
Alteration in immune cell subset phenotype as a long-term response to AP-MODS | 66 months
  Investigating changes to the phenotype of immune cell subsets following an episode of AP; descriptive statistics
Cardiorespiratory dysfunction as a legacy of endothelial injury during AP-MODS | 66 months
  Determination of cardiorespiratory function following AP using physiological measures including cardiopulmonary exercise testing to determine anaerobic threshold. Descriptive measures.

CONTACTS AND LOCATIONS:
Overall Officials: Damian J Mole, MB ChB, Study Director — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sherif AE, McFadyen R, Boyd J, Ventre C, Glenwright M, Walker K, Zheng X, White A, McFadyen L, Connon E, Damaskos D, Steven M, Wackett A, Thomson E, Cameron DC, MacLeod J, Baxter S, Semple S, Morris D, Clark-Stewart S, Graham C, Mole DJ; RESORP research team. Study protocol for resolution of organ injury in acute pancreatitis (RESORP): an observational prospective cohort study. BMJ Open. 2020 Dec 7;10(12):e040200. doi: 10.1136/bmjopen-2020-040200. PMID 33293311
- See also: Protocol publication — http://bmjopen.bmj.com/cgi/content/full/bmjopen-2020-040200